CLINICAL TRIAL: NCT05180552
Title: The HEALiX Trial: Comparing the Efficacy of the HEALiX Device With Wrist Restraints in a Critical Care Setting
Brief Title: The HEALiX: Comparing the Efficacy of the HEALiX Device With Wrist Restraints in a Critical Care Setting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to secure funding or liability insurance
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Eliessa Caplan, Eliessa Caplan, BS, MSN, DNP, RN, CCRN Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TBA2022
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Safety Issues; Device Dislodgement; Device Intolerance; Device Ineffective
Keywords: unplanned extubation; restraints; device removal; critical care unit; patient safety; wrist restraints; sedation; standard of care

STUDY DESIGN:
Intervention Model Description: This randomized control trial will use a quantitative, comparative approach using an experimental and control study group design to measure and compare the outcomes after the subjects are placed in either the HEALiX or wrist restraints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Participants will wear HEALiX Device while intubated and sedated in the critical care setting
  Interventions: Device: HEALiX is an alternative restraint patient safety device
- Control (Active Comparator): Participants will wear wrist restraints while intubated and sedated in the critical care setting
  Interventions: Device: soft wrist restraints

INTERVENTIONS:
Device: HEALiX is an alternative restraint patient safety device — The HEALiX is a rigid, spiral, exoskeleton-like device made of lightweight stainless steel (Austenitic SAE 316 or equivalent) that comes in various sizes to fit different arm lengths circumference of the patient's bicep. After appropriate measuring and following the fit guide, the HEALiX is placed on the patient's arm so that the hand rests on a soft, padded hand cradle. The trajectory of the end hand cradle is at a 30-degree upward angle to prevent peripheral dependent edema. This hand cradle is surrounded by foam to provide increased support for the patient and also to protect the medical team from any injury. A wrist bracelet (wrist assist) goes around the patient's wrist and prevents the patient from removing the device. The spiral exoskeleton holds the arm in a neutral position with contact points with the patient's skin at the upper deltoid region only.
  Arms: Experimental
Device: soft wrist restraints — Soft wrist restraints are padded cloth restraints that are worn by patients on wrist and secured to bed frame.
  Arms: Control

SUMMARY:
The treatment plan for patients requiring mechanical ventilator support is to provide the minimal amount of analgesics and sedatives necessary for the patient to tolerate the ventilator as lower amounts of these drugs has been shown to improve patient outcomes. Patients in this critical state experience confusion, restlessness, and agitation, which sometimes leads to an unplanned removal of a patient's line or medical device. The current standard of care for limiting the movement of mechanically ventilated patients' in the critical care units in hospitals is the use of physical wrist restraints. Researchers demonstrated that wrist restraints are ineffective in preventing the removal of invasive and adjunct devices and have many negative physical, psychological, physiological, and emotional consequences for the patient and their family. In this proposed research, we will use the innovative medical device called the HEALiX, a newly developed device worn on the arms of mechanically ventilated patients that allows freedom of movement and protects from removing adjunct mechanical ventilation devices and invasive monitoring equipment. This randomized controlled trial will investigate the HEALiX device's effectiveness in preventing the removal of invasive monitoring devices (such as endotracheal tubes, central lines, feeding tubes, etc.) compared with the current standard of care, wrist restraints.

DETAILED DESCRIPTION:
This randomized controlled trial's primary purpose is to determine the efficacy of the HEALiX compared with wrist restraints in the adult, intubated patient in the critical care and intermediate care setting. The study's secondary purpose is to understand the acceptability of the HEALiX from healthcare professionals' perspective providing care at the bedside. By recruiting participants for use in the HEALiX RCT study and using the HEALiX with patients during care, the PI will gather information regarding the comparative effectiveness of the HEALiX in a population of critical care patients. This RCT trial will use a quantitative, comparative approach using an experimental and control study group design to measure and compare the outcomes after the subjects are placed in either the HEALiX or wrist restraints.

The setting for the HEALiX Pilot Study will be Penn State Hershey Medical Center in Hershey Pennsylvania. The specific location for the trial will be in several of the academic medical center's critical care units, including Heart and Vascular ICU (HVICU), Surgical Anesthesia ICU (SICU), Neurosurgical Intensive Care Unit (NSICU), and Medical Intensive Care Unit (MICU). Key nursing unit leaders and leaders from other service lines whose clinical input was essential to contribute to this RCT trial's success gave permission to conduct this study.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanically ventilated (with or without tracheostomy)
2. Receiving analgesic-sedating medications
3. Wearing soft wrist restraints
4. Glasgow Coma Scale score > 8
5. Participants must be between ages 18-89 years old
6. English-speaking
7. English speaking legalized authorized representative (LAR)
8. Participants must be admitted under one of the following physician groups: Trauma services or critical care physician group.

Exclusion Criteria:

1. Children (under age 18)
2. Pregnant women
3. Cognitively impaired adults (must be able to follow commands)
4. Prisoners
5. Combative patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2028-08-10 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-09-10 (Estimated)

PRIMARY OUTCOMES:
Unplanned removal of devices | End of intubation (average 7 days)
  Frequency of unplanned removal of lines and self-extubation

SECONDARY OUTCOMES:
Ease of device use | End of intubation (average 7 days)
  Staff perception of ease of HEALiX sizing, application and removal based on Likert scale where 0 is prohibitively hard to use and 5 is extraordinarily easy to use
Days on the ventilator that each patient group remains | End of intubation (average 7 days)
  Days on the ventilator
Number of days in the ICU that each patient group remains | End of ICU stay when patient is transferred to lower level of care (average 10 days)
  Days in ICU
Fentanyl Dosing | 1 Day
  Total Fentanyl dosing in mcg/kg
Propofol Dosing | 1 Day
  Total Propofol dosing in mg/kg
Midazolam Dosing | 1 Day
  Total Midazolam dosing in mg/kg

CONTACTS AND LOCATIONS:
Overall Officials: Eliessa Caplan, DNP, Principal Investigator — Milton S. Hershey Medical Center

IPD SHARING:
Plan to Share IPD: No
Plan to publish in multiple nursing journals and attend research conferences.

REFERENCES:
- [Background] Arumugam S, El-Menyar A, Al-Hassani A, Strandvik G, Asim M, Mekkodithal A, Mudali I, Al-Thani H. Delirium in the Intensive Care Unit. J Emerg Trauma Shock. 2017 Jan-Mar;10(1):37-46. doi: 10.4103/0974-2700.199520. PMID 28243012
- [Background] Balci H, Arslan S. Nurses' Information, Attitude and Practices towards Use of Physical Restraint in Intensive Care Units. J Caring Sci. 2018 Jun 1;7(2):75-81. doi: 10.15171/jcs.2018.012. eCollection 2018 Jun. PMID 29977877
- [Background] Burry L, Rose L, Ricou B. Physical restraint: time to let go. Intensive Care Med. 2018 Aug;44(8):1296-1298. doi: 10.1007/s00134-017-5000-0. Epub 2017 Nov 23. No abstract available. PMID 29170870
- [Background] Jiang H, Li C, Gu Y, He Y. Nurses' perceptions and practice of physical restraint in China. Nurs Ethics. 2015 Sep;22(6):652-60. doi: 10.1177/0969733014557118. Epub 2014 Dec 8. PMID 25488757
- [Background] Johnson K, Curry V, Steubing A, Diana S, McCray A, McFarren A, Domb A. A non-pharmacologic approach to decrease restraint use. Intensive Crit Care Nurs. 2016 Jun;34:12-9. doi: 10.1016/j.iccn.2015.08.004. Epub 2015 Dec 1. PMID 26652790
- [Background] Kwon E, Choi K. Case-control Study on Risk Factors of Unplanned Extubation Based on Patient Safety Model in Critically Ill Patients with Mechanical Ventilation. Asian Nurs Res (Korean Soc Nurs Sci). 2017 Mar;11(1):74-78. doi: 10.1016/j.anr.2017.03.004. Epub 2017 Mar 25. PMID 28388984
- [Background] Lach HW, Leach KM, Butcher HK. Evidence-Based Practice Guideline: Changing the Practice of Physical Restraint Use in Acute Care. J Gerontol Nurs. 2016 Feb;42(2):17-26. doi: 10.3928/00989134-20160113-04. PMID 26820185
- [Background] LeBlanc A, Bourbonnais FF, Harrison D, Tousignant K. The experience of intensive care nurses caring for patients with delirium: A phenomenological study. Intensive Crit Care Nurs. 2018 Feb;44:92-98. doi: 10.1016/j.iccn.2017.09.002. Epub 2017 Oct 6. PMID 28993046
- [Background] Perez D, Peters K, Wilkes L, Murphy G. PHYSICAL RESTRAINTS IN INTENSIVE CARE: EXPERIENCES OF PATIENTS, FAMILIES AND NURSES. Aust Nurs Midwifery J. 2017 May;24(10):45. PMID 29280605
- [Background] Rose L, Dale C, Smith OM, Burry L, Enright G, Fergusson D, Sinha S, Wiesenfeld L, Sinuff T, Mehta S. A mixed-methods systematic review protocol to examine the use of physical restraint with critically ill adults and strategies for minimizing their use. Syst Rev. 2016 Nov 21;5(1):194. doi: 10.1186/s13643-016-0372-8. PMID 27871314
- [Background] Souza LMDS, Santana RF, Capeletto CDSG, Menezes AK, Delvalle R. Factors associated with mechanical restraint in the hospital environment: a cross-sectional study. Rev Esc Enferm USP. 2019 Jun 13;53:e03473. doi: 10.1590/S1980-220X2018007303473. English, Portuguese. PMID 31215614
- [Background] Staggs VS, Olds DM, Cramer E, Shorr RI. Nursing Skill Mix, Nurse Staffing Level, and Physical Restraint Use in US Hospitals: a Longitudinal Study. J Gen Intern Med. 2017 Jan;32(1):35-41. doi: 10.1007/s11606-016-3830-z. Epub 2016 Aug 23. PMID 27553206
- [Background] Ai ZP, Gao XL, Zhao XL. Factors associated with unplanned extubation in the Intensive Care Unit for adult patients: A systematic review and meta-analysis. Intensive Crit Care Nurs. 2018 Aug;47:62-68. doi: 10.1016/j.iccn.2018.03.008. Epub 2018 Apr 10. PMID 29653888